CLINICAL TRIAL: NCT01290094
Title: Interventional, Single Arm, Open Label Study of the Efficacy, Safety and Compliance to the Treatment With Intravenous (IV) Ibandronate (Bonviva®) in the Postmenopausal Osteoporosis Treatment of Bisphosphonates naïve Patients in Daily Practice
Brief Title: A Study of Bonviva/Boniva (Ibandronate) in Biphosphonate-Naïve Women With Post-Menopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25399
Record Dates: First submitted 2011-01-20; First posted 2011-02-04 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-06

CONDITIONS: Post Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 3 mg intravenously every 3 months

SUMMARY:
This single arm, open label study will assess the efficacy and safety of and compliance to treatment with Bonviva/Boniva (ibandronate) in biphosphonate-naïve patients with post-menopausal osteoporosis. Patients will receive Bonviva/Boniva at a dose of 3 mg intravenously every three months. Anticipated time on study treatment is 12 months with a follow-up of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, > 50 years of age
* Diagnosed osteoporosis
* Bone mineral density < minus 2.5 SD or osteoporotic fracture
* At least 3 years after menopause

Exclusion Criteria:

* Impaired renal function
* Contra-indication to Calcium or Vitamin D therapy
* Previous or current treatment with biphosphonates

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Bosnia and Herzegovina (2):
  - Banja Luka
  - Sarajevo

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibandronate: Participants received 3 milligrams (mg) ibandronate via intravenous injection, every 3 months for a total of 12 months (total of 4 injections).
Period: Overall Study
Arm/Group | Ibandronate
Started | 41
Completed | 35
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included participants who received at least 1 dose of study medication and at least 1 efficacy measurement was performed. One participant who was enrolled in the study initially, withdrew informed consent and was excluded from ITT population.
Groups:
- Ibandronate: Participants received 3 mg ibandronate via intravenous injection, every 3 months for a total of 12 months (total of 4 injections).
Arm/Group | Ibandronate
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.60 (5.812)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Mean Lumbar Spine Bone Mineral Density (BMD) at Month 12
Description: Percent change was calculated as [(measure at time "t" minus [-] measure at baseline) divided by (/) measure at baseline] multiplied by (*) 100, where t=12 months. The baseline value is used as a reference to calculate the relative change from baseline.
Time Frame: Baseline, Month 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate
Number analyzed (Participants) | 40
percent change | 5.67 (7.86)
Statistical Analysis 1: Comparison: Ibandronate; Test type: Superiority or Other; p < 0.0005, Paired t-test — P-value for percent change from baseline was from a paired samples t-test

2. Primary Outcome: Percent Change From Baseline in Mean Lumbar Spine BMD at Month 24
Description: Percent change was calculated as [(measure at time "t" - measure at baseline)/measure at baseline]*100, where t=24 months. The baseline value is used as a reference to calculate the relative change from baseline.
Time Frame: Baseline, Month 24
Population: ITT population. Here "number of participants analyzed" included participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate
Number analyzed (Participants) | 35
percent change | 5.27 (8.00)
Statistical Analysis 1: Comparison: Ibandronate; Test type: Superiority or Other; p < 0.0005, Paired t-test — P-value for percent change from baseline was from a paired samples t-test

3. Primary Outcome: Percent Change From Baseline in Mean Hip Bone BMD at Month 12
Description: Percent change was calculated as [(measure at time "t" - measure at baseline)/measure at baseline]*100, where t=12 months. The baseline value is used as a reference to calculate the relative change from baseline.
Time Frame: Baseline, Month 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate
Number analyzed (Participants) | 40
percent change | 2.68 (4.66)
Statistical Analysis 1: Comparison: Ibandronate; Test type: Superiority or Other; p = 0.001, Paired t-test — P-value for percent change from baseline was from a paired samples t-test

4. Primary Outcome: Percent Change From Baseline in Mean Hip BMD at Month 24
Description: as for outcome 2
Time Frame: Baseline, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate
Number analyzed (Participants) | 35
percent change | 1.71 (5.09)
Statistical Analysis 1: Comparison: Ibandronate; Test type: Superiority or Other; p = 0.056, Paired t-test — P-value for percent change from baseline was from a paired samples t-test

5. Secondary Outcome: Percent Change From Baseline in Lumbar Spine T-score at Month 12 and 24
Description: Percent change was calculated as [(measure at time "t" - measure at baseline)/measure at baseline]*100, where t=12 and 24 months. The baseline value is used as a reference to calculate the relative change from baseline. T-score is the number of standard deviations above or below the mean for a healthy 30 year old adult of the same sex and ethnicity as the participant. A T-score with above -1 is normal bone density level. A T-score between -1 and -2.5 means that the bone density is below normal and it might be a sign of an osteopenia and may also lead into osteoporosis. A T-score below -2.5 indicates osteoporosis. A T-score below -2.5 in combination with a prevalent fracture indicates serious osteoporosis.
Time Frame: Baseline, Month 12, Month 24
Population: ITT population. Here "n" included participants who were evaluable at specified time point for the given arm.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate
Number analyzed (Participants) | 40
percent change
  Change at Month 12 (n=40) | 13.47 (12.23)
  Change at Month 24 (n=35) | 12.48 (13.43)
Statistical Analysis 1: Comparison: Ibandronate; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test — Month 12: P-value for percent change from baseline was from a Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Ibandronate; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test — Month 24: P-value for percent change from baseline was from a Wilcoxon signed rank test

6. Secondary Outcome: Percent Change From Baseline in Total Hip T-score at Month 12 and 24
Description: as for outcome 5
Time Frame: Baseline, Month 12, Month 24
Population: ITT population. Here "n" included participants who were evaluable at specified time point for the given arm.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate
Number analyzed (Participants) | 40
percent change
  Change at Month 12 (n=40) | 9.31 (16.75)
  Change at Month 24 (n=35) | 5.98 (17.90)
Statistical Analysis 1: Comparison: Ibandronate; Test type: Superiority or Other; p < 0.0005, Paired t-test — Month 12: P-value for percent change from baseline was from a paired samples t-test
Statistical Analysis 2: Comparison: Ibandronate; Test type: Superiority or Other; p = 0.027, Paired t-test — Month 24: P-value for percent change from baseline was from a paired samples t-test

7. Secondary Outcome: Percentage of Participants Who Received All Planned Study Medication (Compliance)
Time Frame: Baseline up to Month 12
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Ibandronate
Number analyzed (Participants) | 40
percentage of participants | 100

8. Secondary Outcome: Correlation Coefficient of Participant's Profile With Compliance
Description: Participant's profile included age, year since menopause, fracture history, and BMD at baseline.
Time Frame: Baseline up to Month 12
Population: ITT population.
Measure: Number; unit: correlation coefficient
Arm/Group | Ibandronate
Number analyzed (Participants) | 40
correlation coefficient | NA — Since there was 100% compliance, it was decided not to perform the analysis of correlation coefficient of participant's Profile With Compliance.

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up (Month 24)
Description: ITT population.
Groups:
- Ibandronate: Participants received 3 mg ibandronate via intravenous injection, every 3 months for 9 months (total of 4 injections).
Arm/Group | Ibandronate
Serious Adverse Events (participants affected / at risk) | 9/40
Other Adverse Events (participants affected / at risk) | 20/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=40)
Fractures (Injury, poisoning and procedural complications) | 3
Eyelid disorder (Eye disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Loss of conciousness (Nervous system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Gallbladder disorder (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate (N=40)
Gastrointestinal pain (Gastrointestinal disorders) | 2
Flu like symptoms (General disorders) | 12
Injection site reaction (General disorders) | 2
Neuralgia (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.